CLINICAL TRIAL: NCT01263691
Title: A Parallel-arm, Double-blind, Randomized, Placebo-controlled, Dose-ranging Clinical Trial Evaluating the Safety, Tolerability and Immunogenicity of AV7909 in Healthy Adults
Brief Title: Safety, Tolerability and Immunogenicity Study of AV7909 Anthrax Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EBS.AVA.201 / DMID 10-0013; HHSN272200800051C (Other Grant/Funding Number: BARDA/NIAID)
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Bacillus Anthracis (Anthrax) Infection
Keywords: AVA; AV7909; Anthrax vaccine
MeSH Terms: conditions — Anthrax; Infections | interventions — Biothrax; Anthrax Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- BioThrax (Active Comparator): BioThrax, 0.5 mL AVA per dose
  Interventions: Biological: BioThrax
- AV7909 Formulation 1 (Experimental): 0.5 mL AVA + 0.5 mg CPG 7909 per 0.5 mL dose
  Interventions: Biological: AV7909 Formulation 1
- AV7909 Formulation 2 (Experimental): 0.5 mL AVA + 0.25 mg CPG 7909 per 0.5 mL dose
  Interventions: Biological: AV7909 Formulation 2
- AV7909 Formulation 3 (Experimental): 0.25 mL AVA + 0.5 mg CPG 7909 per 0.5 mL dose
  Interventions: Biological: AV7909 Formulation 3
- AV7909 Formulation 4 (Experimental): 0.25 mL AVA + 0.25 mg CPG 7909 per 0.5 mL dose
  Interventions: Biological: AV7909 Formulation 4
- Control (Placebo Comparator): Saline control
  Interventions: Drug: Control

INTERVENTIONS:
Biological: BioThrax — BioThrax
  Other Names: Anthrax Vaccine Adsorbed (AVA)
  Arms: BioThrax
Biological: AV7909 Formulation 1 — AV7909 Formulation 1
  Arms: AV7909 Formulation 1
Biological: AV7909 Formulation 2 — AV7909 Formulation 2
  Arms: AV7909 Formulation 2
Biological: AV7909 Formulation 3 — AV7909 Formulation 3
  Arms: AV7909 Formulation 3
Biological: AV7909 Formulation 4 — AV7909 Formulation 4
  Arms: AV7909 Formulation 4
Drug: Control — Saline control
  Arms: Control

SUMMARY:
The purpose of this Phase 1 clinical trial is to evaluate the safety, tolerability, and immunogenicity of AV7909 anthrax vaccine in healthy adults. In this study, healthy male and female subjects between 18 and 50 years of age will receive vaccinations via the intramuscular (IM) route at Days 0 and 14. Safety and tolerability will be evaluated via laboratory tests, physical examinations, vital signs, adverse events (AEs), concomitant medications, and local and systemic signs and symptoms of reactogenicity.

DETAILED DESCRIPTION:
AV7909 is a new vaccine which is a combination of BioThrax (also called anthrax vaccine, adsorbed or AVA), a FDA-licensed vaccine, and CPG 7909. CPG 7909 is a synthetic short DNA sequence that has been shown to be an effective vaccine adjuvant, and one which increases the speed and the degree of the immune response to Protective Antigen (PA), the major vaccine antigen. In the current study, the safety, tolerability, and antibody response to PA will be studied for four different combinations of AVA and CPG 7909, and compared to both AVA and a saline placebo. All formulations of AV7909 have the same or less AVA than the licensed AVA vaccine and all have less CPG 7909 per dose than the formulation used in the first Phase I volunteer study of CPG 7909 combined with AVA.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 50 years of age, inclusive, at the time of enrollment.
* Be in good health as determined by the investigator from medical history and a physical examination.
* If a pre-menopausal female, must be using acceptable methods of birth control.
* Have all hematology and chemistry parameters (measured at Screening) within the laboratory's normal range.
* Have negative values for the following tests at Screening: Hepatitis C antibody, anti-Human Immunodeficiency Virus (Anti-HIV-1/-2/-O), and anti-Hepatitis B Core Antigen (Anti-HBc).
* Be willing and capable of complying with all aspects of the protocol through completion of the required visits.
* Have not donated blood in the preceding 8 weeks and are willing to not donate blood or plasma within 56 days after dosing.
* Have adequate venous access for repeat phlebotomies.
* Have read, understood and signed an informed consent form.

Exclusion Criteria:

Key Exclusion Criteria:

* A known anaphylactic response, severe systematic response, or serious hypersensitivity reaction to a prior immunization.
* Prior immunization with anthrax vaccine, recombinant Protective Antigen (rPA) vaccine, or known exposure to anthrax organisms.
* Have previously served in the military or plans to enlist in the military from Screening through Day 84.
* Have participated in anthrax therapeutic or vaccine trials (monoclonal anti-protective antigen (PA) or anthrax immune globulins or anthrax vaccines).
* Participation in any investigational clinical trial within 30 days preceding the Screening visit or planning to participate in a clinical trial requiring dosing through the Day 194 visit.
* A history of drug or alcohol abuse within 12 months prior to Screening, or a positive result on a urine drug screen for amphetamines, barbiturates, benzodiazepines, cocaine, marijuana, methylenedioxymethamphetamine opiates, oxycodone, phencyclidine, propoxyphene, or tricyclic antidepressants.
* Blood pressure greater than 145 millimeters of mercury (mmHg) systolic or 90 mmHg diastolic.
* Past history of significant autoimmune disease such as rheumatoid arthritis, lupus erythematous, psoriasis, glomerulonephritis, or autoimmune thyroiditis.
* A medical condition that, in the opinion of the Principal Investigator (PI), could adversely impact the subject's participation, safety, or conduct of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bernton, MD, Study Director — Emergent Biosolutions, Inc.
Locations (3):
- United States (3):
  - Miami Research Associates, Miami, Florida
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Result] Hopkins RJ, Daczkowski NF, Kaptur PE, Muse D, Sheldon E, LaForce C, Sari S, Rudge TL, Bernton E. Randomized, double-blind, placebo-controlled, safety and immunogenicity study of 4 formulations of Anthrax Vaccine Adsorbed plus CPG 7909 (AV7909) in healthy adult volunteers. Vaccine. 2013 Jun 26;31(30):3051-8. doi: 10.1016/j.vaccine.2013.04.063. Epub 2013 May 10. PMID 23701746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 27 December 2010 to 08 March 2012 at three medical centers in the U.S.
Pre-assignment Details: All 105 enrolled participants who met inclusion and exclusion criteria were dosed.
Groups:
- BioThrax: Participants between 18 and 50 years of age who received two doses of BioThrax (0.5 mL) intramuscularly (IM) on Days 0 and 14
- AV7909 Formulation 1: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 1 (0.5 mL anthrax vaccine adsorbed [AVA] + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- AV7909 Formulation 2: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 2 (0.5 mL anthrax vaccine adsorbed [AVA] + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- AV7909 Formulation 3: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 3 (0.25 mL anthrax vaccine adsorbed [AVA] + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- AV7909 Formulation 4: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 4 (0.25 mL anthrax vaccine adsorbed [AVA] + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- Saline: Participants between 18 and 50 years of age who received two doses of saline placebo (0.5 mL) IM on Days 0 and 14
Period: Overall Study
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Started | 18 | 18 | 17 | 19 | 18 | 15
Completed | 15 | 18 | 16 | 18 | 18 | 15
Not Completed | 3 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AV7909 Formulation 1: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 1 (0.5 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- AV7909 Formulation 2: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 2 (0.5 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- AV7909 Formulation 3: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 3 (0.25 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- AV7909 Formulation 4: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 4 (0.25 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14
- Total: Total of all reporting groups
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline | Total
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 1 | 0 | 0 | 5
  Between 18 and 65 years | 17 | 17 | 15 | 18 | 18 | 15 | 100
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (9.27) | 32.8 (10.31) | 32.4 (10.75) | 32.6 (9.15) | 31.4 (10.72) | 31.4 (8.61) | 32.0 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 9 | 8 | 9 | 7 | 51
  Male | 9 | 9 | 8 | 11 | 9 | 8 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 6 | 6 | 3 | 3 | 25
  Not Hispanic or Latino | 14 | 15 | 11 | 13 | 15 | 12 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 6 | 3 | 2 | 15
  White | 15 | 17 | 15 | 12 | 15 | 13 | 87
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 17 | 19 | 18 | 15 | 105
Weight [Mean (Standard Deviation); unit: kilograms] | 80.06 (18.799) | 83.99 (16.137) | 75.75 (12.232) | 78.39 (19.021) | 76.24 (15.649) | 79.74 (23.140) | 79.03 (17.487)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Injection Site Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the First Vaccination (Day 0)
Description: Subjects recorded solicited injection site reactions (ISRs) (redness, swelling, tenderness, pain, itching, arm motion limitation) on diary cards for 7 days following the first injection (Day 0).
  All local reactions collected by subjects on diary cards were recorded as adverse events.
  Severity of ISR was assessed using a grading scale based on FDA Guidance "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials."
  Swelling/edema and redness/erythema were graded by the greater of two perpendicular measurements of diameter rated as follows:
  * Grade 0: none
  * Grade 1: <3 cm
  * Grade 2: 3 to 10 cm
  * Grade 3: >10 cm
  For all other ISRs, the following scale was used:
  * Grade 0: not present
  * Grade 1: present with no limitation of activity
  * Grade 2: interfering with daily activities or requiring non-narcotic treatment
  * Grade 3: preventing normal daily activities or requiring narcotic analgesia
Time Frame: Days 0-6
Measure: Number; unit: Participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
Participants
  Any Injection Site Reaction | 11 | 17 | 13 | 12 | 16 | 1
  Grade 1 Injection Site Reaction | 9 | 9 | 11 | 6 | 11 | 1
  Grade 2 Injection Site Reaction | 1 | 6 | 2 | 6 | 5 | 0
  Grade 3 Injection Site Reaction | 1 | 2 | 0 | 0 | 0 | 0
  Any Redness | 0 | 2 | 1 | 2 | 1 | 0
  Grade 1 Redness | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Redness | 0 | 1 | 1 | 2 | 1 | 0
  Any Swelling | 1 | 4 | 1 | 1 | 2 | 0
  Grade 1 Swelling | 0 | 0 | 1 | 0 | 1 | 0
  Grade 2 Swelling | 0 | 2 | 0 | 1 | 1 | 0
  Grade 3 Swelling | 1 | 2 | 0 | 0 | 0 | 0
  Any Tenderness | 10 | 16 | 11 | 11 | 13 | 1
  Grade 1 Tenderness | 9 | 13 | 10 | 10 | 11 | 1
  Grade 2 Tenderness | 1 | 3 | 1 | 1 | 2 | 0
  Any Injection Site Pain | 5 | 14 | 12 | 8 | 11 | 0
  Grade 1 Injection Site Pain | 4 | 12 | 12 | 7 | 8 | 0
  Grade 2 Injection Site Pain | 1 | 2 | 0 | 1 | 3 | 0
  Any Injection Site Itching | 0 | 2 | 2 | 0 | 0 | 0
  Grade 1 Injection Site Itching | 0 | 1 | 2 | 0 | 0 | 0
  Grade 2 Injection Site Itching | 0 | 1 | 0 | 0 | 0 | 0
  Any Arm Motion Limitation | 8 | 13 | 8 | 9 | 10 | 0
  Grade 1 Arm Motion Limitation | 7 | 8 | 7 | 4 | 6 | 0
  Grade 2 Arm Motion Limitation | 1 | 5 | 1 | 5 | 4 | 0

2. Secondary Outcome: Peak TNA NF50 GMT for All Subjects in the Immunogenicity Population and by Gender After IM Administration of Investigational Product on Days 0 and 14.
Description: Toxin neutralizing antibody (TNA) levels in blinded serum samples were measured using a validated anthrax lethal toxin neutralization assay. The primary assay endpoint was the 50% neutralization factor (TNA NF50). TNA NF50 is calculated as the ratio of the 50% effective dose (ED50) of the test sample to the ED50 of a reference serum. Values below the lower limit of quantitation (LLOQ) of the assay (ED50 of 33) were replaced with one-half the LLOQ (ED50 of 16.5) for calculation of geometric mean titer (GMT) and statistical analysis. GMT is based on log transformation.
Time Frame: Day 0 (pre-dose), 7, 14 (pre-dose), 21, 28, 35, 42, 56, 70, and 84.
Population: Participants 18 and 50 years of age who received two doses of saline placebo (0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- BioThrax: Participants between 18 and 50 years of age who received two doses of BioThrax (0.5 mL) intramuscularly (IM) on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- AV7909 Formulation 1: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 1 (0.5 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- AV7909 Formulation 2: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 2 (0.5 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- AV7909 Formulation 3: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 3 (0.25 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- AV7909 Formulation 4: Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 4 (0.25 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Saline: Participants between 18 and 50 years of age who received two doses of saline placebo (0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male BioThrax: Male Participants between 18 and 50 years of age who received two doses of BioThrax (0.5 mL) intramuscularly (IM) on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male AV7909 Formulation 1: Male Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 1 (0.5 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male AV7909 Formulation 2: Male Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 2 (0.5 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male AV7909 Formulation 3: Male Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 3 (0.25 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male AV7909 Formulation 4: Male Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 4 (0.25 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male Saline: Male Participants between 18 and 50 years of age who received two doses of saline placebo (0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female BioThrax: Female Participants between 18 and 50 years of age who received two doses of BioThrax (0.5 mL) intramuscularly (IM) on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female AV7909 Formulation 1: Female Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 1 (0.5 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female AV7909 Formulation 2: Female Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 2 (0.5 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female AV7909 Formulation 3: Female Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 3 (0.25 mL AVA + 0.5 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female AV7909 Formulation 4: Female Participants between 18 and 50 years of age who received two doses of AV7909 Formulation 4 (0.25 mL AVA + 0.25 mg CPG 7909; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female Saline: Female Participants between 18 and 50 years of age who received two doses of saline placebo (0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline | Male BioThrax | Male AV7909 Formulation 1 | Male AV7909 Formulation 2 | Male AV7909 Formulation 3 | Male AV7909 Formulation 4 | Male Saline | Female BioThrax | Female AV7909 Formulation 1 | Female AV7909 Formulation 2 | Female AV7909 Formulation 3 | Female AV7909 Formulation 4 | Female Saline
Number analyzed (Participants) | 16 | 17 | 16 | 18 | 18 | 15 | 8 | 9 | 8 | 8 | 9 | 7 | 8 | 8 | 8 | 10 | 9 | 8
geometric mean titer | 0.15 [0.07 to 0.30] | 3.40 [2.33 to 4.94] | 4.02 [2.46 to 6.57] | 2.81 [1.50 to 5.26] | 1.93 [0.85 to 4.43] | 0.04 [0.02 to 0.08] | 0.19 [0.06 to 0.62] | 3.44 [1.84 to 6.43] | 4.19 [2.19 to 7.98] | 2.99 [1.32 to 6.78] | 2.45 [0.54 to 11.12] | 0.03 [NA to NA] — All values were equal and below the lower limit of quantitation | 0.11 [0.04 to 0.36] | 3.35 [1.91 to 5.88] | 3.87 [1.54 to 9.71] | 2.68 [0.92 to 7.80] | 1.53 [0.53 to 4.39] | 0.06 [0.01 to 0.21]

3. Primary Outcome: Percentage of Subjects With Injection Site Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the First Vaccination (Day 0)
Description: as for outcome 1
Time Frame: Days 0-6
Measure: Number; unit: Percentage of Participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
Percentage of Participants
  Any Injection Site Reaction | 61.1 | 94.4 | 76.5 | 63.2 | 88.9 | 6.7
  Grade 1 Injection Site Reaction | 50.0 | 50.0 | 64.7 | 31.6 | 61.1 | 6.7
  Grade 2 Injection Site Reaction | 5.6 | 33.3 | 11.8 | 31.6 | 27.8 | 0
  Grade 3 Injection Site Reaction | 5.6 | 11.1 | 0 | 0 | 0 | 0
  Any Redness | 0 | 11.1 | 5.9 | 10.5 | 5.6 | 0
  Grade 1 Redness | 0 | 5.6 | 0 | 0 | 0 | 0
  Grade 2 Redness | 0 | 5.6 | 5.9 | 10.5 | 5.6 | 0
  Any Swelling | 5.6 | 22.2 | 5.9 | 5.3 | 11.1 | 0
  Grade 1 Swelling | 0 | 0 | 5.9 | 0 | 5.6 | 0
  Grade 2 Swelling | 0 | 11.1 | 0 | 5.3 | 5.6 | 0
  Grade 3 Swelling | 5.6 | 11.1 | 0 | 0 | 0 | 0
  Any Tenderness | 55.6 | 88.9 | 64.7 | 57.9 | 72.2 | 6.7
  Grade 1 Tenderness | 50.0 | 72.2 | 58.8 | 52.6 | 61.1 | 6.7
  Grade 2 Tenderness | 5.6 | 16.7 | 5.9 | 5.3 | 11.1 | 0
  Any Injection Site Pain | 27.8 | 77.8 | 70.6 | 42.1 | 61.1 | 0
  Grade 1 Injection Site Pain | 22.2 | 66.7 | 70.6 | 36.8 | 44.4 | 0
  Grade 2 Injection Site Pain | 5.6 | 11.1 | 0 | 5.3 | 16.7 | 0
  Any Injection Site Itching | 0 | 11.1 | 11.8 | 0 | 0 | 0
  Grade 1 Injection Site Itching | 0 | 5.6 | 11.8 | 0 | 0 | 0
  Grade 2 Injection Site Itching | 0 | 5.6 | 0 | 0 | 0 | 0
  Any Arm Motion Limitation | 44.4 | 72.2 | 47.1 | 47.4 | 55.6 | 0
  Grade 1 Arm Motion Limitation | 38.9 | 44.4 | 41.2 | 21.1 | 33.3 | 0
  Grade 2 Arm Motion Limitation | 5.6 | 27.8 | 5.9 | 26.3 | 22.2 | 0

4. Primary Outcome: Incidence of Injection Site Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the Second Vaccination (Day 14)
Description: Subjects recorded solicited injection site reactions (ISRs) (redness, swelling, tenderness, pain, itching, arm motion limitation) on diary cards for 7 days following the second injection (Day 14).
  All local reactions collected by subjects on diary cards were recorded as adverse events.
  Severity of ISR was assessed using a grading scale based on FDA Guidance "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials."
  Swelling/edema and redness/erythema were graded by the greater of two perpendicular measurements of diameter rated as follows:
  * Grade 0: none
  * Grade 1: <3 cm
  * Grade 2: 3 to 10 cm
  * Grade 3: >10 cm
  For all other ISRs, the following scale was used:
  * Grade 0: not present
  * Grade 1: present with no limitation of activity
  * Grade 2: interfering with daily activities or requiring non-narcotic treatment
  * Grade 3: preventing normal daily activities or requiring narcotic analgesia
Time Frame: Days 14-20
Measure: Number; unit: Participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
Participants
  Any Injection Site Reaction | 11 | 16 | 12 | 11 | 13 | 0
  Grade 1 Injection Site Reaction | 6 | 8 | 9 | 6 | 7 | 0
  Grade 2 Injection Site Reaction | 4 | 6 | 3 | 3 | 6 | 0
  Grade 3 Injection Site Reaction | 1 | 2 | 0 | 2 | 0 | 0
  Any Redness | 1 | 3 | 2 | 3 | 0 | 0
  Grade 1 Redness | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Redness | 1 | 3 | 2 | 2 | 0 | 0
  Grade 3 Redness | 0 | 0 | 0 | 1 | 0 | 0
  Any Swelling | 2 | 4 | 2 | 2 | 1 | 0
  Grade 1 Swelling | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Swelling | 2 | 3 | 2 | 2 | 0 | 0
  Grade 3 Swelling | 0 | 1 | 0 | 0 | 0 | 0
  Any Tenderness | 11 | 13 | 11 | 10 | 12 | 0
  Grade 1 Tenderness | 8 | 8 | 11 | 8 | 9 | 0
  Grade 2 Tenderness | 2 | 5 | 0 | 2 | 3 | 0
  Grade 3 Tenderness | 1 | 0 | 0 | 0 | 0 | 0
  Any Injection Site Pain | 6 | 13 | 10 | 8 | 6 | 0
  Grade 1 Injection Site Pain | 2 | 10 | 10 | 6 | 3 | 0
  Grade 2 Injection Site Pain | 3 | 2 | 0 | 2 | 3 | 0
  Grade 3 Injection Site Pain | 1 | 1 | 0 | 0 | 0 | 0
  Any Injection Site Itching | 2 | 3 | 3 | 2 | 0 | 0
  Grade 1 Injection Site Itching | 2 | 2 | 3 | 2 | 0 | 0
  Grade 3 Injection Site Itching | 0 | 1 | 0 | 0 | 0 | 0
  Any Arm Motion Limitation | 8 | 11 | 7 | 8 | 8 | 0
  Grade 1 Arm Motion Limitation | 4 | 6 | 6 | 4 | 3 | 0
  Grade 2 Arm Motion Limitation | 3 | 4 | 1 | 3 | 5 | 0
  Grade 3 Arm Motion Limitation | 1 | 1 | 0 | 1 | 0 | 0

5. Primary Outcome: Percentage of Subjects With Injection Site Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the Second Vaccination (Day 14)
Description: as for outcome 4
Time Frame: Days 14-20
Measure: Number; unit: Percentage of Participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
Percentage of Participants
  Any Injection Site Reaction | 61.1 | 88.9 | 70.6 | 57.9 | 72.2 | 0
  Grade 1 Injection Site Reaction | 33.3 | 44.4 | 52.9 | 31.6 | 38.9 | 0
  Grade 2 Injection Site Reaction | 22.2 | 33.3 | 17.6 | 15.8 | 33.3 | 0
  Grade 3 Injection Site Reaction | 5.6 | 11.1 | 0 | 10.5 | 0 | 0
  Any Redness | 5.6 | 16.7 | 11.8 | 15.8 | 0 | 0
  Grade 2 Redness | 5.6 | 16.7 | 11.8 | 10.5 | 0 | 0
  Grade 3 Redness | 0 | 0 | 0 | 5.3 | 0 | 0
  Any Swelling | 11.1 | 22.2 | 11.8 | 10.5 | 5.6 | 0
  Grade 1 Swelling | 0 | 0 | 0 | 0 | 5.6 | 0
  Grade 2 Swelling | 11.1 | 16.7 | 11.8 | 10.5 | 0 | 0
  Grade 3 Swelling | 0 | 5.6 | 0 | 0 | 0 | 0
  Any Tenderness | 61.1 | 72.2 | 64.7 | 52.6 | 66.7 | 0
  Grade 1 Tenderness | 44.4 | 44.14 | 64.7 | 42.1 | 50.0 | 0
  Grade 2 Tenderness | 11.1 | 27.8 | 0 | 10.5 | 16.7 | 0
  Grade 3 Tenderness | 5.6 | 0 | 0 | 0 | 0 | 0
  Any Injection Site Pain | 33.3 | 72.2 | 58.8 | 42.1 | 33.3 | 0
  Grade 1 Injection Site Pain | 11.1 | 55.6 | 58.8 | 31.6 | 16.7 | 0
  Grade 2 Injection Site Pain | 16.7 | 11.1 | 0 | 10.5 | 16.7 | 0
  Grade 3 Injection Site Pain | 5.6 | 5.6 | 0 | 0 | 0 | 0
  Any Injection Site Itching | 11.1 | 16.7 | 17.6 | 10.5 | 0 | 0
  Grade 1 Injection Site Itching | 11.1 | 11.1 | 17.6 | 10.5 | 0 | 0
  Grade 3 Injection Site Itching | 0 | 5.6 | 0 | 0 | 0 | 0
  Any Arm Motion Limitation | 44.4 | 61.1 | 41.2 | 42.1 | 44.4 | 0
  Grade 1 Arm Motion Limitation | 22.2 | 33.3 | 35.3 | 21.1 | 16.7 | 0
  Grade 2 Arm Motion Limitation | 16.7 | 22.2 | 5.9 | 15.8 | 27.8 | 0
  Grade 3 Arm Motion Limitation | 5.6 | 5.6 | 0 | 5.3 | 0 | 0

6. Primary Outcome: Incidence of Systemic Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the First Injection (Day 0)
Description: Subjects recorded solicited systemic reactions (fever, fatigue, muscle aching, headache, nausea/GI upset) on diary cards for 7 days following each of two injections (Days 0 and 14) All systemic reactions collected by subjects on diary cards were recorded as adverse events.
  Severity of systemic reactions was assessed using a grading scale based on FDA Guidance titled "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials."
  Toxicity grades for fever were derived from body temperature using the following scale:
  * Grade 0: <100°F
  * Grade 1: 100.0 - 101.5°F
  * Grade 2: 101.6 - 102.9°F ;
  * Grade 3: 103.0 - 105.0°F
  For all other systemic reactions, the following scale was used:
  * Grade 0: not present
  * Grade 1: present with no limitation of activity
  * Grade 2: interfering with daily activities or requiring non-narcotic treatment
  * Grade 3: preventing normal daily activities or requiring narcotic analgesia
Time Frame: Days 0-6
Measure: Number; unit: Participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
Participants
  Any Systemic Reaction | 10 | 12 | 7 | 3 | 7 | 5
  Grade 1 Systemic Reaction | 8 | 5 | 5 | 3 | 2 | 4
  Grade 2 Systemic Reaction | 2 | 7 | 2 | 0 | 4 | 1
  Grade 3 Systemic Reaction | 0 | 0 | 0 | 0 | 1 | 0
  Any Fever | 0 | 2 | 1 | 0 | 0 | 2
  Grade 1 Fever | 0 | 2 | 1 | 0 | 0 | 2
  Any Fatigue | 6 | 9 | 3 | 3 | 4 | 2
  Grade 1 Fatigue | 5 | 4 | 1 | 3 | 2 | 2
  Grade 2 Fatigue | 1 | 5 | 2 | 0 | 2 | 0
  Any Muscle Ache | 4 | 8 | 3 | 0 | 2 | 2
  Grade 1 Muscle Ache | 4 | 6 | 1 | 0 | 2 | 1
  Grade 2 Muscle Ache | 0 | 2 | 2 | 0 | 0 | 1
  Any Headache | 6 | 11 | 5 | 1 | 5 | 2
  Grade 1 Headache | 6 | 4 | 3 | 1 | 1 | 1
  Grade 2 Headache | 0 | 7 | 2 | 0 | 3 | 1
  Grade 3 Headache | 0 | 0 | 0 | 0 | 1 | 0
  Any Nausea / GI Upset | 1 | 4 | 2 | 2 | 2 | 2
  Grade 1 Nausea / GI Upset | 0 | 1 | 2 | 2 | 2 | 1
  Grade 2 Nausea / GI Upset | 1 | 3 | 0 | 0 | 0 | 1

7. Primary Outcome: Percentage of Subjects With Systemic Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the First Injection (Day 0)
Description: as for outcome 6
Time Frame: Days 0-6
Measure: Number; unit: percentage of participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
percentage of participants
  Any Systemic Reaction | 55.6 | 66.7 | 41.2 | 15.8 | 38.9 | 33.3
  Grade 1 Systemic Reaction | 44.4 | 27.8 | 29.4 | 15.8 | 11.1 | 26.7
  Grade 2 Systemic Reactions | 11.1 | 38.9 | 11.8 | 0 | 22.2 | 6.7
  Grade 3 Systemic Reaction | 0 | 0 | 0 | 0 | 5.6 | 0
  Any Fever | 0 | 11.1 | 5.9 | 0 | 0 | 13.3
  Grade 1 Fever | 0 | 11.1 | 5.9 | 0 | 0 | 13.3
  Any Fatigue | 33.3 | 50.0 | 17.6 | 15.8 | 22.2 | 13.3
  Grade 1 Fatigue | 27.8 | 22.2 | 5.9 | 15.8 | 11.1 | 13.3
  Grade 2 Fatigue | 5.6 | 27.8 | 11.8 | 0 | 11.1 | 0
  Any Muscle Ache | 22.2 | 44.4 | 17.6 | 0 | 11.1 | 13.3
  Grade 1 Muscle Ache | 22.2 | 33.3 | 5.9 | 0 | 11.1 | 6.7
  Grade 2 Muscle Ache | 0 | 11.1 | 11.8 | 0 | 0 | 6.7
  Any Headache | 33.3 | 61.1 | 29.4 | 5.3 | 27.8 | 13.3
  Grade 1 Headache | 33.3 | 22.2 | 17.6 | 5.3 | 5.6 | 6.7
  Grade 2 Headache | 0 | 8.9 | 11.8 | 0 | 16.47 | 6.7
  Grade 3 Headache | 0 | 0 | 0 | 0 | 5.6 | 0
  Any Nausea / GI Upset | 5.6 | 22.2 | 11.8 | 10.5 | 11.1 | 13.3
  Grade 1 Nausea / GI Upset | 0 | 5.6 | 11.8 | 10.5 | 11.1 | 6.7
  Grade 2 Nausea / GI Upset | 5.6 | 16.7 | 0 | 0 | 0 | 6.7

8. Primary Outcome: Incidence of Systemic Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the Second Injection (Day 14)
Description: as for outcome 6
Time Frame: Days 14-20
Measure: Number; unit: participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
participants
  Any Systemic Reaction | 7 | 14 | 7 | 4 | 9 | 2
  Grade 1 Systemic Reaction | 3 | 8 | 6 | 2 | 4 | 1
  Grade 2 Systemic Reactions | 3 | 5 | 1 | 2 | 5 | 1
  Grade 3 Systemic Reaction | 1 | 1 | 0 | 0 | 0 | 0
  Any Fever | 0 | 0 | 0 | 0 | 1 | 0
  Grade 1 Fever | 0 | 0 | 0 | 0 | 1 | 0
  Any Fatigue | 4 | 8 | 4 | 3 | 7 | 1
  Grade 1 Fatigue | 3 | 5 | 3 | 1 | 4 | 1
  Grade 2 Fatigue | 1 | 2 | 1 | 2 | 3 | 0
  Grade 3 Fatigue | 0 | 1 | 0 | 0 | 0 | 0
  Any Muscle Ache | 5 | 9 | 3 | 2 | 7 | 0
  Grade 1 Muscle Ache | 3 | 5 | 2 | 1 | 4 | 0
  Grade 2 Muscle Ache | 1 | 3 | 1 | 1 | 3 | 0
  Grade 3 Muscle Ache | 1 | 1 | 0 | 0 | 0 | 0
  Any Headache | 5 | 7 | 3 | 3 | 7 | 1
  Grade 1 Headache | 2 | 5 | 3 | 2 | 3 | 0
  Grade 2 Headache | 2 | 2 | 0 | 1 | 4 | 1
  Grade 3 Headache | 1 | 0 | 0 | 0 | 0 | 0
  Any Nausea / GI Upset | 1 | 3 | 0 | 0 | 3 | 0
  Grade 1 Nausea / GI Upset | 1 | 2 | 0 | 0 | 2 | 0
  Grade 2 Nausea / GI Upset | 0 | 1 | 0 | 0 | 1 | 0

9. Primary Outcome: Percentage of Subjects With Systemic Reactions From Subject Diary Cards by Injection and Severity (Mild, Moderate or Severe) Following the Second Injection (Day 14)
Description: as for outcome 6
Time Frame: Days 14-20
Measure: Number; unit: percentage of participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
percentage of participants
  Any Systemic Reaction | 38.9 | 77.8 | 41.2 | 21.1 | 50.0 | 13.3
  Grade 1 Systemic Reaction | 16.7 | 44.14 | 35.3 | 10.5 | 22.2 | 6.7
  Grade 2 Systemic Reactions | 16.7 | 27.8 | 5.9 | 10.5 | 27.8 | 6.7
  Grade 3 Systemic Reaction | 5.6 | 5.6 | 0 | 0 | 0 | 0
  Any Fever | 0 | 0 | 0 | 0 | 5.6 | 0
  Grade 1 Fever | 0 | 0 | 0 | 0 | 5.6 | 0
  Any Fatigue | 22.2 | 44.4 | 23.5 | 15.8 | 38.9 | 6.7
  Grade 1 Fatigue | 16.7 | 27.8 | 17.6 | 5.3 | 22.2 | 6.7
  Grade 2 Fatigue | 5.6 | 11.1 | 5.9 | 10.5 | 16.7 | 0
  Grade 3 Fatigue | 0 | 5.6 | 0 | 0 | 0 | 0
  Any Muscle Ache | 27.8 | 50.0 | 17.6 | 10.5 | 38.9 | 0
  Grade 1 Muscle Ache | 16.7 | 27.8 | 11.8 | 5.3 | 22.2 | 0
  Grade 2 Muscle Ache | 5.6 | 16.7 | 5.9 | 5.3 | 16.7 | 0
  Grade 3 Muscle Ache | 5.6 | 5.6 | 0 | 0 | 0 | 0
  Any Headache | 27.8 | 38.9 | 17.6 | 15.8 | 38.9 | 6.7
  Grade 1 Headache | 11.1 | 27.8 | 17.6 | 10.5 | 16.7 | 0
  Grade 2 Headache | 11.1 | 11.1 | 0 | 5.3 | 22.2 | 6.7
  Grade 3 Headache | 5.6 | 0 | 0 | 0 | 0 | 0
  Any Nausea / GI Upset | 5.6 | 16.7 | 0 | 0 | 16.7 | 0
  Grade 1 Nausea / GI Upset | 5.6 | 11.1 | 0 | 0 | 11.1 | 0
  Grade 2 Nausea / GI Upset | 0 | 5.6 | 0 | 0 | 5.6 | 0

10. Primary Outcome: Incidence of Hematology, Serum Chemistry, and Urinalysis Abnormalities Reported as Adverse Events
Description: Hematology test included hemoglobin, hematocrit, white blood cell count, absolute lymphocyte count, absolute neutrophil count, absolute eosinophil count, and platelet count. Serum chemistry test included albumin, alkaline phosphatase, total bilirubin, blood urea nitrogen, creatinine, glucose, calcium, potassium, alanine aminotransferase, aspartate aminotransferase, and lactate dehydrogenase. Urinalysis included appearance, color, pH, specific gravity, ketones, protein, glucose, bilirubin, nitrite, urobilinogen, and occult blood.
  Hematology tests were done on Days 0, 1, 2, 7, 28, and 56. Serum chemistry tests and urinalysis were done on Days 0, 7, 28, and 56.
Time Frame: Days 0-56
Measure: Number; unit: participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
participants
  Alanine aminotransferase increased | 0 | 0 | 1 | 0 | 1 | 1
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 2 | 0
  Blood creatinine increased | 0 | 0 | 1 | 0 | 0 | 0
  Blood lactate dehydrogenase increased | 0 | 0 | 0 | 0 | 0 | 1
  Blood urea increased | 0 | 1 | 0 | 0 | 0 | 0
  Hepatic enzyme increased | 0 | 0 | 0 | 0 | 0 | 1
  Hyperkalemia | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 1 | 0 | 2 | 0 | 0
  Hypokalemia | 0 | 0 | 1 | 1 | 0 | 0
  Hypomagnesemia | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocyte count decreased | 0 | 6 | 3 | 1 | 4 | 0
  Neutropenia | 1 | 1 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 1 | 0 | 0 | 0 | 0
  Protein urine | 0 | 1 | 0 | 1 | 1 | 1
  Red blood cells urine positive | 0 | 0 | 1 | 0 | 0 | 0
  White blood cell count decreased | 2 | 5 | 4 | 0 | 2 | 1
  White blood cell count increased | 0 | 1 | 0 | 0 | 0 | 0
  White blood cells urine positive | 0 | 0 | 1 | 0 | 0 | 0

11. Primary Outcome: Percentage of Subjects With Hematology, Serum Chemistry, and Urinalysis Abnormalities Reported as Adverse Events
Description: as for outcome 10
Time Frame: Days 0-56
Measure: Number; unit: percentage of participants
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 18 | 15
percentage of participants
  Alanine aminotransferase increased | 0 | 0 | 5.9 | 0 | 5.6 | 6.7
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 11.1 | 0
  Blood creatinine increased | 0 | 0 | 5.9 | 0 | 0 | 0
  Blood lactate dehydrogenase increased | 0 | 0 | 0 | 0 | 0 | 6.7
  Blood urea increased | 0 | 5.6 | 0 | 0 | 0 | 0
  Hepatic enzyme increased | 0 | 0 | 0 | 0 | 0 | 6.7
  Hyperkalemia | 0 | 5.6 | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 5.6 | 0 | 10.5 | 0 | 0
  Hypokalemia | 0 | 0 | 5.9 | 5.3 | 0 | 0
  Hypomagnesemia | 0 | 0 | 0 | 5.3 | 0 | 0
  Lymphocyte count decreased | 0 | 33.3 | 17.6 | 5.3 | 22.2 | 0
  Neutropenia | 5.6 | 5.6 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 5.6 | 0 | 0 | 0 | 0
  Protein urine | 0 | 5.6 | 0 | 5.3 | 5.6 | 6.7
  Red blood cells urine positive | 0 | 0 | 5.9 | 0 | 0 | 0
  White blood cell count decreased | 11.1 | 27.8 | 23.5 | 0 | 11.1 | 6.7
  White blood cell count increased | 0 | 5.6 | 0 | 0 | 0 | 0
  White blood cells urine positive | 0 | 0 | 5.9 | 0 | 0 | 0

12. Secondary Outcome: Median Time to Peak TNA NF50 GMT for All Subjects in the Immunogenicity Population and by Gender After IM Administration of Investigational Product on Days 0 and 14.
Description: Toxin neutralizing antibody (TNA) levels in blinded serum samples were measured using a validated anthrax lethal toxin neutralization assay. The primary assay endpoint was the 50% neutralization factor (TNA NF50). TNA NF50 is calculated as the ratio of the 50% effective dose (ED50) of the test sample to the ED50 of a reference serum. Values below the LLOQ of the assay (ED50 of 33) were replaced with one-half the LLOQ (ED50 of 16.5) for calculation of geometric mean titer (GMT) and statistical analysis. GMT is based on log transformation.
Time Frame: Day 0 (pre-dose), 7, 14 (pre-dose), 21, 28, 35, 42, 56, 70, and 84.
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Groups:
- Saline: Participants between 18 and 50 years of age who received two doses of saline; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Male Saline: Male participants between 18 and 50 years of age who received two doses of saline; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
- Female Saline: Female participants between 18 and 50 years of age who received two doses of saline; total volume 0.5 mL) IM on Days 0 and 14 Antibody titers were assessed in the immunogenicity population, which included subjects who received both vaccinations, had immunogenicity data within the allowable window, and had no protocol violations that could affect TNA values (n=100).
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline | Male BioThrax | Male AV7909 Formulation 1 | Male AV7909 Formulation 2 | Male AV7909 Formulation 3 | Male AV7909 Formulation 4 | Male Saline | Female BioThrax | Female AV7909 Formulation 1 | Female AV7909 Formulation 2 | Female AV7909 Formulation 3 | Female AV7909 Formulation 4 | Female Saline
Number analyzed (Participants) | 16 | 17 | 16 | 18 | 18 | 15 | 8 | 9 | 8 | 8 | 9 | 7 | 8 | 8 | 8 | 10 | 9 | 8
days | 28.0 [7 to 42] | 29.0 [21 to 42] | 28.0 [22 to 35] | 28.5 [27 to 42] | 29.0 [7 to 42] | 7.0 [6 to 70] | 28.0 [7 to 35] | 28.0 [21 to 42] | 28.0 [22 to 35] | 28.0 [28 to 39] | 28.0 [7 to 35] | 7.0 [7 to 8] | 18.5 [7 to 42] | 32.0 [28 to 36] | 28.0 [22 to 30] | 29.0 [27 to 42] | 35.0 [21 to 42] | 7.0 [6 to 70]

13. Secondary Outcome: TNA NF50 GMTs Across Study Days After IM Administration of Investigational Product on Days 0 and 14.
Description: as for outcome 12
Time Frame: Day 0 (pre-dose), 7, 14 (pre-dose), 21, 28, 35, 42, 56, 70, and 84.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Number analyzed (Participants) | 16 | 17 | 16 | 18 | 18 | 15
geometric mean titer
  Day 0 | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 7 | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 14 | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.03 [NA to NA] — All values were below the LLOQ for the assay | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.05] | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 21 | 0.04 [0.0276 to 0.0651] | 1.27 [0.78 to 2.07] | 0.77 [0.32 to 1.83] | 0.90 [0.46 to 1.75] | 0.44 [0.17 to 1.10] | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 28 | 0.13 [0.06 to 0.28] | 3.05 [2.07 to 4.52] | 3.85 [2.40 to 6.20] | 2.54 [1.26 to 5.12] | 1.73 [0.77 to 3.89] | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 35 | 0.15 [0.07 to 0.32] | 2.61 [1.82 to 3.75] | 2.89 [1.80 to 4.61] | 2.23 [1.11 to 4.45] | 1.56 [0.68 to 3.59] | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 42 | 0.13 [0.07 to 0.24] | 2.01 [1.37 to 2.95] | 2.03 [1.32 to 3.12] | 1.78 [0.95 to 3.34] | 1.17 [0.53 to 2.59] | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 56 | 0.09 [0.05 to 0.16] | 1.18 [0.81 to 1.71] | 1.52 [0.97 to 2.36] | 1.09 [0.58 to 2.07] | 0.76 [0.37 to 1.61] | 0.03 [NA to NA] — All values were below the LLOQ for the assay
  Day 70 | 0.06 [0.04 to 0.10] | 0.85 [0.56 to 1.29] | 0.91 [0.58 to 1.41] | 0.71 [0.40 to 1.25] | 0.55 [0.26 to 1.16] | 0.04 [0.02 to 0.08]
  Day 84 | 0.05 [0.04 to 0.08] | 0.67 [0.42 to 1.08] | 0.69 [0.44 to 1.10] | 0.55 [0.32 to 0.94] | 0.39 [0.20 to 0.77] | 0.03 [NA to NA] — All values were below the LLOQ for the assay

ADVERSE EVENTS:
Time Frame: Serious adverse event data were collected at study visits from Day 0 to Day 84 and during safety follow-up telephone calls at 6 and 12 months.
Description: Serious adverse events were coded using Medical Dictionary for Regulatory Activities (MedDRA®) Version 14.0.
  Severity of laboratory toxicities were assessed using the Toxicity Grading Scale in the protocol.
  For determination of Other Adverse Events frequency, all study Arms were combined.
Arm/Group | BioThrax | AV7909 Formulation 1 | AV7909 Formulation 2 | AV7909 Formulation 3 | AV7909 Formulation 4 | Saline
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/18 | 1/17 | 0/19 | 0/18 | 1/15
Other Adverse Events (participants affected / at risk) | 16/18 | 18/18 | 14/17 | 14/19 | 18/18 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioThrax (N=18) | AV7909 Formulation 1 (N=18) | AV7909 Formulation 2 (N=17) | AV7909 Formulation 3 (N=19) | AV7909 Formulation 4 (N=18) | Saline (N=15)
Elevated hepatic enzymes (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Elevated hepatic enzymes (Grade 4 elevated Alanine aminotransferase [ALT], Grade 3 elevated Aspartate aminotransferase [AST]) on Day 28 was attributed to an acute Epstein-Barr infection (unrelated to vaccination).
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Glioblastoma multiforme was reported during 6-month safety follow-up telephone call. The event was assessed as unrelated to vaccination.
Death (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Road traffic accident resulting in death was reported during 12-month safety follow-up telephone call. The event was assessed as unrelated to vaccination.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioThrax (N=18) | AV7909 Formulation 1 (N=18) | AV7909 Formulation 2 (N=17) | AV7909 Formulation 3 (N=19) | AV7909 Formulation 4 (N=18) | Saline (N=15)
Fatigue (General disorders) | 8 (13) | 13 (21) | 6 (14) | 4 (6) | 9 (13) | 3 (4)
Headache (Nervous system disorders) | 6 (15) | 11 (20) | 5 (9) | 5 (5) | 10 (17) | 2 (6)
Injection Site Reaction (General disorders) | 15 (27) | 18 (36) | 14 (27) | 14 (24) | 16 (32) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 6 (6) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (12) | 10 (21) | 4 (11) | 2 (2) | 10 (14) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (14) | 3 (3) | 2 (2) | 4 (5) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (7) | 1 (1) | 3 (6) | 1 (2) | 2 (2) | 2 (3)
White Blood Cell Count Decreased (Investigations) | 2 (3) | 5 (5) | 4 (5) | 0 (0) | 2 (3) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sternal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 1 (1) | 1 (1) | 0 | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor is responsible for public disclosure of study data. Any proposed publication is subject to review agreed between National Institute of Allergy and Infectious Disease (NIAID) and Emergent; between Emergent and the contract research organizations (CROs)/vendors; and between the CROs and the site Principal Investigator. Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.